CLINICAL TRIAL: NCT03776370
Title: A Clinical Cohort Study on the Effect of Preserving Left Colonic Artery During Radical Resection of Rectal Cancer on Anastomotic Leakage and Oncology Efficacy
Brief Title: Preserving Left Colonic Artery During Radical Resection of Rectal Cancer
Status: Completed | Type: Observational
Sponsor: Third Military Medical University (Other)
Responsible Party: Principal Investigator, Weidong Tong, Clinical Professor, Third Military Medical University
Other Study IDs: 20181155
Record Dates: First submitted 2018-12-09; First posted 2018-12-14 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Postoperative Complications; Proteinosis
Keywords: rectal cancer; Postoperative Complications; Preserve the left colonic artery
MeSH Terms: conditions — Postoperative Complications; Rectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preserve the left colonic artery: Preservation of left colonic artery in rectal cancer surgery.
  Interventions: Procedure: Preserve the left colonic artery
- The left colonic artery is not preserved: The left colonic artery was dissected in rectal cancer surgery
  Interventions: Procedure: The left colonic artery is not preserved

INTERVENTIONS:
Procedure: Preserve the left colonic artery — Preservation of left colonic artery in rectal cancer surgery.
  Groups: Preserve the left colonic artery
Procedure: The left colonic artery is not preserved — The left colonic artery was dissected in rectal cancer surgery.
  Groups: The left colonic artery is not preserved

SUMMARY:
To evaluate the feasibility and clinical significance of preserving left colonic artery in rectal cancer surgery.The investigators will focus on the effect of preserving left colonic artery during radical resection of rectal cancer on anastomotic leakage and oncology efficacy.

DETAILED DESCRIPTION:
The investigators performed three-dimensional (3D) reconstruction to investigate the vascular anatomy, including the inferior mesenteric artery (IMA) and left colic artery (LCA),to help make pre-operative strategies of rectal cancer surgery.The investigators will preserving the left colonic artery during rectal cancer surgery and evaluate its feasibility and clinical significance.The investigators will focus on the effect of preserving left colonic artery during radical resection of rectal cancer on anastomotic leakage and oncology efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Pathological biopsy confirmed adenocarcinoma of the rectum；
2. Preoperative assessment of tolerance to surgery without major organ dysfunction；
3. Patients must be able to understand and voluntarily sign written informed consent；
4. The surgical method is laparoscopic or robotic anterior rectal cancer resection.

Exclusion Criteria:

1. The patient cannot tolerate the operation；
2. Refusal to sign informed consent；
3. Patients with distant metastasis of rectal cancer；
4. The surgical method was changed to miles or Hartman;
5. Unable to complete the follow - up

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who underwent laparoscopic or robotic anterior rectal resections carried out by two surgeons at Daping Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-01-01 (Actual)

PRIMARY OUTCOMES:
The incidence of postoperative anastomotic leakage was compared between the two groups. | Within 30 days after surgery
  The incidence of anastomotic leakage within 30 days after surgery was compared between the intervention group and the control group.
The distant metastasis rates of rectal cancer between the two groups were compared. | Two years after surgery
  The incidence of distant metastasis rectal cancer within two years after surgery was compared between the intervention group and the control group.
The local recurrence rates of rectal cancer between the two groups were compared. | Two years after surgery
  The incidence of local recurrence rectal cancer within two years after surgery was compared between the intervention group and the control group.
The five-year survival rates of rectal cancer between the two groups were compared. | Five years after surgery
  The 5-year survival rates of rectal cancer in the intervention group and the control group were compared.

CONTACTS AND LOCATIONS:
Overall Officials: Wei d tong, PhD, Principal Investigator — Army Military Medical University
Locations (2):
- China (2):
  - zongming,Kang, Chongqing, Chongqing Municipality
  - zongming,Kang, Yuzhong, Chongqing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Fan YC, Ning FL, Zhang CD, Dai DQ. Preservation versus non-preservation of left colic artery in sigmoid and rectal cancer surgery: A meta-analysis. Int J Surg. 2018 Apr;52:269-277. doi: 10.1016/j.ijsu.2018.02.054. Epub 2018 Mar 1. PMID 29501795
- [Result] Sekimoto M, Takemasa I, Mizushima T, Ikeda M, Yamamoto H, Doki Y, Mori M. Laparoscopic lymph node dissection around the inferior mesenteric artery with preservation of the left colic artery. Surg Endosc. 2011 Mar;25(3):861-6. doi: 10.1007/s00464-010-1284-7. Epub 2010 Aug 20. PMID 20725744
- [Derived] Zheng H, Li F, Xie X, Zhao S, Huang B, Tong W. Preservation versus nonpreservation of the left colic artery in anterior resection for rectal cancer: a propensity score-matched analysis. BMC Surg. 2022 May 10;22(1):164. doi: 10.1186/s12893-022-01614-y. PMID 35538516